CLINICAL TRIAL: NCT06357741
Title: Clinical Study of Desuzumab in the Treatment of Knee Osteoarthritis
Acronym: CSODITTOKO
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tian Hongtao, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: 202286
Record Dates: First submitted 2023-08-05; First posted 2024-04-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: denosumab; knee osteoarthritis; curative effect
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Denosumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some patients receiving denosumab injections requested to withdraw from the trial to undergo knee replacement, during which synovial tissue samples were collected for H&E, IHC staining, and Western blot. Knee replacement inherently requires partial synovectomy to prevent postoperative joint crepitus and alleviate inflammatory pain. The resected pathological tissues during knee replacement-including synovium and cartilage-are routinely sent for pathological examination to exclude neoplasms or infections, confirm diagnoses, and guide postoperative management. Studies suggest that denosumab may effectively reduce periprosthetic fracture risk. Thus, even after trial withdrawal, patients can benefit from its osteoporotic therapeutic effects in preventing post-arthroplasty complications such as prosthetic loosening and periprosthetic fractures. In addition, we could also check whether there are some protective effects by denosumab on molecular level.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- desumumab1: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab2: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 3: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab4: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab5: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 6: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab7: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 8: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 9: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 10: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 11: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 12: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 13: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 14: 60mg, single injection.
  Interventions: Drug: Denosumab
- desumumab 15: 60mg, single injection.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Desumumab, 60mg single injection

SUMMARY:
As an activator of inhibiting nuclear factor kB receptor, denosumab affects osteoclast differentiation and development by inhibiting OPG/RANKL-RANK bone regulatory axis pathway. Therefore, denosumab is widely used in the treatment of bone diseases such as osteoporosis. Osteoporosis is closely related to knee osteoarthritis. RANKL-RANK pathway also plays a key role in the pathogenesis of knee osteoarthritis. Therefore, the investigators propose the hypothesis that denosumab can effectively treat knee osteoarthritis.

DETAILED DESCRIPTION:
basic overview at present, about 60% of the elderly over 60 years old in China suffer from knee osteoarthritis, and there are more than 100million patients with knee osteoarthritis in China. It is estimated that the world's elderly population will reach 2.02 billion in 2050, and China will reach 480million, accounting for almost 5% of the global elderly population, making it the country with the largest elderly population in the world . At present, the treatment of knee osteoarthritis is only analgesic drugs to alleviate symptoms, and there is no effective treatment to reverse the progress of knee osteoarthritis. Therefore, many patients with knee osteoarthritis eventually face knee replacement surgery. In 2019, there were nearly 400000 knee replacement operations in China, and the number will increase by 30% next year, which is undoubtedly a huge economic expenditure for patients. Denosumab is widely used in the treatment of osteoporosis by inhibiting nuclear factor kB activating factor (rank). Rank and RANKL are important molecular systems that regulate bone remodeling and the dynamic balance of bone metabolism. In osteoporosis, the combination of rank and RANKL will directly promote the differentiation and maturation of osteoblasts, enhance their bone resorption activity and prevent their apoptosis. The relative transcription of rank in osteoclasts and their precursor cells is significantly increased, which promotes bone loss and leads to osteoporosis. RANKL-RANK pathway also plays a key role in the pathogenesis of osteoarthritis . The chondrocytes and synovial cells of patients with knee osteoarthritis will produce interleukin-1 after being stimulated by trauma, wear and tear β （IL-1 β）、 TNF- α And prostaglandin E2 (PGE2) and other inflammatory factors promote osteoclasts to secrete metalloproteinases (MMPs) and matrix protease tissue inhibitors (TIMPs), and these inflammatory factors can directly stimulate RANKL to induce the production of osteoclasts, resulting in the destruction of cartilage matrix, the impairment of bone regeneration ability, the irreversible degradation of cartilage tissue, and even apoptosis . At the same time, it has been reported in the literature that osteoporosis and knee osteoarthritis are closely related, and the two promote each other, forming a vicious circle . The symptoms of knee osteoarthritis can be relieved by treating osteoporosis. However, there is no report about denosumab in the treatment of knee osteoarthritis. Therefore, this project plans to use a prospective, single center randomized controlled trial to study the clinical efficacy of denosumab in the treatment of patients with knee osteoarthritis and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with knee osteoarthritis whose inclusion criteria meet the "diagnostic criteria for arthritis" .
* no drug contraindications .
* aged between 45 and 75 .
* committed to follow the research procedures, And cooperate with the •implementation of the whole process study .
* the patient understands the relevant treatment process .
* the patient has the ability to give informed consent .
* The patient had not recently taken any medication that affected observation.
* the subjects must meet all the inclusion criteria to be eligible to participate in the study .

Exclusion Criteria:

* mental illness .
* patients with malignant tumors.
* patients with other infectious diseases .
* patients with metabolic bone disease, diabetes and hyperthyroidism.
* patients who cannot actively cooperate in the treatment.
* hypocalcemia.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subject recruitment
  * the research object comes from outpatient patients
  * recruitment advertisement for publicity
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee pain relief | 1,3,6 months
  OKS function of knee joint at 1,3 and 6 months, VAS pain score at 1,3 and 6 months;

SECONDARY OUTCOMES:
Knee pain relief and incidence of adverse reactions | 1,3,6 months
  Knee joint WOMAC score（maximum：250 ，minimum：0） at 1,3 and 6 months；incidence of adverse reactions;EQ-5D quality of life score at 1,3 and 6 months；

CONTACTS AND LOCATIONS:
Overall Officials: Tian Hongtao, Doctorate, Principal Investigator — Wuhan Union Medical College Hospital
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] He XF, Zhang L, Zhang CH, Zhao CR, Li H, Zhang LF, Tian GF, Guo MF, Dai Z, Sui FG. Berberine alleviates oxidative stress in rats with osteoporosis through receptor activator of NF-kB/receptor activator of NF-kB ligand/osteoprotegerin (RANK/RANKL/OPG) pathway. Bosn J Basic Med Sci. 2017 Nov 20;17(4):295-301. doi: 10.17305/bjbms.2017.2596. PMID 29055350
- [Background] Ernest TL, Kondrashov PE. The role of excessive body weight and meniscal instability in the progression of osteoarthritis in a rat model. Knee. 2018 Dec;25(6):1151-1156. doi: 10.1016/j.knee.2018.07.009. Epub 2018 Aug 13. PMID 30115587
- [Background] Zhou J, Liao Y, Zeng Y, Xie H, Fu C, Li N. Effect of intervention initiation timing of pulsed electromagnetic field on ovariectomy-induced osteoporosis in rats. Bioelectromagnetics. 2017 Sep;38(6):456-465. doi: 10.1002/bem.22059. Epub 2017 May 16. PMID 28510268
- [Result] Sobacchi C, Frattini A, Guerrini MM, Abinun M, Pangrazio A, Susani L, Bredius R, Mancini G, Cant A, Bishop N, Grabowski P, Del Fattore A, Messina C, Errigo G, Coxon FP, Scott DI, Teti A, Rogers MJ, Vezzoni P, Villa A, Helfrich MH. Osteoclast-poor human osteopetrosis due to mutations in the gene encoding RANKL. Nat Genet. 2007 Aug;39(8):960-2. doi: 10.1038/ng2076. Epub 2007 Jul 15. PMID 17632511

DOCUMENTS (1):
  • Study Protocol (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT06357741/Prot_001.pdf